CLINICAL TRIAL: NCT05916313
Title: A Phase Ib Open-label, Multi-center, Dose Escalation Trial of BI 764532 Given as Monotherapy Administered by Repeated Intravenous Infusions in Patients With Glioma Expressing DLL3
Brief Title: A Study to Test How Well Different Doses of BI 764532 Are Tolerated by People With a Tumour in the Brain That is Positive for DLL3
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0003; U1111-1290-7234 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP)); 2022-501766-22-01 (EU CTIS Number)
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BI 764532, dose escalation cohort (Experimental)
  Interventions: Drug: BI 764532

INTERVENTIONS:
Drug: BI 764532 — BI 764532
  Other Names: Obrixtamig

SUMMARY:
This study (1438-0003) is open to adults with a tumour in the brain that is positive for the tumour marker delta-like 3 (DLL3). This study is in people with advanced cancer for whom previous treatment was not successful.

The purpose of this study is to find out the highest dose of BI 764532 that people with a brain tumour that is positive for DLL3 can tolerate. BI 764532 is an antibody-like molecule that can attach and link together the cancer cells and T-cells of the immune system (DLL3/CD3 bispecific). This may help the immune system fight cancer.

Participants get BI 764532 infusions into a vein when starting treatment. If there is benefit for the participants and if they can tolerate it, the treatment is continued. During this time, participants visit the study site at regular intervals. The total number of visits depends on how they respond to and tolerate the treatment. The first study visits include staying to monitor participants' safety. Doctors record any unwanted effects and regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years old and at least at the legal age of consent in countries where it is greater than 18 years at the time of signature of the first informed consent form (ICF1).
2. Signed and dated written informed consent (ICF1 and ICF2) in accordance with International Council for Harmonisation-Good clinical practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Patients with histologically confirmed primary progressive diffuse glioma who have failed standard of care therapies.
4. Availability of archival tumour tissue for Delta-like 3 (DLL3) expression by central assessment.
5. Tumours must be positive for DLL3 expression by immunohistochemistry (IHC) on archived tumour tissue according to central pathology review.
6. Documented unequivocal progression after radiotherapy and/or chemotherapy with measurable disease by response assessment in neuro-oncology (RANO) criteria.
7. Karnofsky performance score ≥70. Further inclusion criteria apply.

Exclusion Criteria:

1. Previous treatment in this trial.
2. Current enrolment in another investigational device or drug trial.
3. Presence of extracranial metastatic or leptomeningeal disease.
4. Previous treatment with therapies targeting DLL3.
5. Prior treatment with bevacizumab or other anti-vascular endothelial growth factor (anti-VEGF) or anti-angiogenic treatment within 6 months prior to first administration of BI 764532.
6. Recent anti-cancer therapy: treatment with any other anticancer drug within 21 days or within 5 half-life periods (whichever is shorter) prior to first administration of BI 764532.
7. Radiotherapy within the 3 months prior to the diagnosis of progression; unless tumour progression is clearly outside the radiation field or tumour progression is unequivocally proven by surgery/biopsy.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT) during the maximum tolerated dose (MTD) evaluation period | up to 4 weeks

SECONDARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT) during the entire treatment period | up to 26 months

CONTACTS AND LOCATIONS:
Locations (12):
- United States (2):
  - University of California Irvine, Orange, California
  - SCRI Oncology Partners, Nashville, Tennessee
- Salzburg Cancer Research Institute, Salzburg, Austria
- Germany (3):
  - Universitätsklinikum Frankfurt, Frankfurt
  - Klinikum der Universität München AÖR, München
  - Universitätsklinikum Tübingen, Tübingen
- Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam, Netherlands
- Spain (2):
  - Hospital del Mar, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Cantonal Hospital of Aarau, Aarau
  - University Hospital of Lausanne, Lausanne
  - University Hosp. Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com